CLINICAL TRIAL: NCT07287254
Title: The Effect of Different Types of Music on Pain and Anxiety During Wound Care Procedures in Patients With Venous Ulcers: A Randomized Controlled Trial
Brief Title: The Effect of Different Types of Music on Pain and Anxiety During Wound Care Procedures in Patients With Venous Ulcers
Acronym: MUPAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Gülay OYUR ÇELİK, Asst. Prof. Dr., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0553
Record Dates: First submitted 2025-11-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Venous Leg Ulcer; Pain; Anxiety
Keywords: Music Therapy; Pain; Anxiety; Venous Leg Ulcer; Wound Dressing; Nursing Intervention
MeSH Terms: conditions — Varicose Ulcer; Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Turkish music (Experimental): Music Intervention
  Interventions: Other: Turkish Music Intervention
- Western music (Experimental): Music Intervention
  Interventions: Other: Western Music Intervention
- control group (No Intervention): control group

INTERVENTIONS:
Other: Turkish Music Intervention — The music intervention was prepared by a music therapy specialist. Patients in the intervention groups listened only to the music portion of the therapy via a USB player. The music was played continuously and repeatedly in the outpatient clinic for approximately 30-60 minutes (for patients whose dressing lasted at least 30-45 minutes) at a moderate volume of 20-45 dB (sufficient to avoid interfering with speech or communication). To enhance the effectiveness of music therapy, the listening experience was structured with gradual variations in tempo and dynamics. Major tonal sequences were preferred to stimulate neural activity. The selected pieces included instrumental Western Classical music and Turkish music (Nihavend makam), starting at a tempo of 60 bpm (Adagio) and gradually increasing to 100 bpm (Andante). Examples include W.A. Mozart's Flute and Horn Concertos for Western Classical music, and instrumental compositions in the Nihavend makam for Turkish music.
  Other Names: music therapy
  Arms: Turkish music
Other: Western Music Intervention — The music intervention was prepared by a music therapy specialist. Patients in the intervention groups listened only to the music portion of the therapy via a USB player. The music was played continuously and repeatedly in the outpatient clinic for approximately 30-60 minutes (for patients whose dressing lasted at least 30-45 minutes) at a moderate volume of 20-45 dB (sufficient to avoid interfering with speech or communication).[22] To enhance the effectiveness of music therapy, the listening experience was structured with gradual variations in tempo and dynamics. Major tonal sequences were preferred to stimulate neural activity. The selected pieces included instrumental Western Classical music and Turkish music (Nihavend makam), starting at a tempo of 60 bpm (Adagio) and gradually increasing to 100 bpm (Andante). Examples include W.A. Mozart's Flute and Horn Concertos for Western Classical music, and instrumental compositions in the Nihavend makam for Turkish music.
  Other Names: Music therapy
  Arms: Western music

SUMMARY:
Objective: To evaluate the effects of different types of music (instrumental Turkish music and Western music without lyrics) played during wound care on pain, anxiety, and patient satisfaction among individuals with venous ulcers.

Methods: In this randomized controlled trial, 97 patients with venous ulcers were assigned to three groups: Western Music (n=32), Turkish Music (n=32), and Control (n=33). Patients in the music groups listened to their assigned music during routine wound dressing, while all patients received individualized, evidence-based care. Pain and anxiety were measured with VAS and STAI before, during, and after dressing, and patient satisfaction was assessed with VAS post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the outpatient clinic with venous leg ulcers (CEAP classification: C6 - active ulcers)
* Age between 18 and 65 years
* Absence of neuropathy
* Willingness to listen to music and voluntary participation
* Literacy (able to read and write)
* No visual or hearing impairments
* No cognitive deficits; fully oriented to time, place, and person
* Turkish-speaking
* No formal music education

Exclusion Criteria:

* Diagnosis of diabetes or diabetic foot
* Use of analgesic medications prior to or during routine wound care
* Individuals younger than 18 or older than 65 years
* Patients with psychiatric disorders
* Individuals with intellectual disabilities
* Patients with severe anxiety levels (STAI-S score 60-79 indicating severe anxiety)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by the Visual Analog Scale (VAS) | Immediately before wound dressing; Periprocedural period; Immediately after wound dressing
  Pain intensity will be assessed using a 0-10 cm Visual Analog Scale (VAS), where higher scores indicate more severe pain.
State anxiety level measured by the State Anxiety Inventory (STAI-S) score | Before the wound dressing procedure; Immediately after the wound dressing procedure
  State anxiety will be assessed using the State Anxiety Inventory (STAI-S), a 20-item validated self-report scale that measures situational (state) anxiety. Scores range from 20 to 80, with higher scores indicating greater anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi Üniversitesi, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary outcome results will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year and ending 2 years after the publication of results
Access Criteria: Data will be made available upon reasonable request to the corresponding author. Requests must include a research proposal and will be reviewed for scientific merit and ethical compatibility.